CLINICAL TRIAL: NCT04183725
Title: Reduning Injection for the Treatment of Influenza in Children:a Randomized, Double-blinded, Parallel-controlled Clinical Study
Brief Title: Clinical Study of Reduning Injection for the Treatment of Influenza in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Children's Hospital of Soochow University (Other); Anhui Provincial Children's Hospital (Other); Qilu Children's Hospital of Shandong University (Other); Tianjin 4th Centre Hospital (Unknown); Renmin Hospital of Wuhan University (Other); Hebei Maternity&Child Healthcare Hospital (Unknown); The Second Affiliated Hospital of Jiaxing University (Other); Hunan University of Traditional Chinese Medicine (Other); Affiliated Hospital of Shanxi University of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reduning injection
Record Dates: First submitted 2019-11-22; First posted 2019-12-03 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Influenza in Children
Keywords: Reduning injection; efficacy and safety; time of temperature recovery; randomized; double blind; parallel control; multi-center clinical study
MeSH Terms: interventions — reduning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Reduning injection +Oseltamivir phosphate granule simulants
  Interventions: Drug: Reduning injection
- Control group (Active Comparator): Oseltamivir phosphate granules+ Reduning injection simulants
  Interventions: Drug: Oseltamivir phosphate granules

INTERVENTIONS:
Drug: Reduning injection — Reduning injection:
  2≤Age≤5,0.5ml/kg/day,<10ml/day+5％GS/0.9％NS 50～100ml,iv drip 30～40gtt/min qd*5; 6≤Age≤10,10ml/day+5％GS/0.9％NS 100～200ml,iv drip 30～60gtt/min qd*5; 11≤Age≤13,15ml/day+5％GS/0.9％NS 200～250ml,iv drip 30～60gtt/min qd*5; Age=14,20ml/day+5％GS/0.9％NS 250ml,iv drip 30～60gtt/min qd*5.
  Oseltamivir phosphate granules simulants:
  Weight≤15kg,30mg,po,bid*5; 15<Weight≤23kg,45mg,po,bid*5; 23<Weight≤40kg,60mg,po,bid*5; Weight>40kg,75mg,po,bid*5.
  Other Names: Oseltamivir phosphate granule simulants
  Arms: Experimental group
Drug: Oseltamivir phosphate granules — Oseltamivir phosphate granules:
  Weight≤15kg,30mg,po,bid*5; 15<Weight≤23kg,45mg,po,bid*5; 23<Weight≤40kg,60mg,po,bid*5; Weight>40kg,75mg,po,bid*5.
  +Reduning injection simulants: 2≤Age≤5,0.5ml/kg/day,<10ml/day+5％GS/0.9％NS 50～100ml,iv drip 30～40gtt/min qd*5; 6≤Age≤10,10ml/day+5％GS/0.9％NS 100～200ml,iv drip 30～60gtt/min qd*5; 11≤Age≤13,15ml/day+5％GS/0.9％NS 200～250ml,iv drip 30～60gtt/min qd*5; Age=14,20ml/day+5％GS/0.9％NS 250ml,iv drip 30～60gtt/min qd*5.
  Other Names: Reduning injection simulants
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety of Reduning injection for the treatment of influenza in children.

DETAILED DESCRIPTION:
The clinical efficacy of Traditional Chinese Medicine(TCM) injection was verified by evaluating the efficacy and safety of Reduning injection in the treatment of influenza in children, so as to provide more therapeutic programs for the treatment of influenza in children and provide clinical research evidence for clinical medication.In this study, a parallel control, randomized, double-blind,multi-center trial will be used to design the optimal efficacy of positive drugs.The time of body temperature that return normal was taken as the main therapeutic index.According to the formula of mean superiority test,the number of sample was calculated to 240 cases, with 120 cases in each experimental group and control group.The experimental group was treated with Reduning injection and Oseltamivir phosphate granule simulants, while the control group was treated with Oseltamivir phosphate granules and Reduning injection simulants .Each group will be treated for 5 days.Primary outcome measure this study was mainly from one dimension:Time of temperature recovery.Secondary outcome measures include the time when the fever begins to subside,the time of disease to alleviate,the degree of disease remission,disappearance rate of individual symptoms, etc.Before and after treatment,the temperature of each group was observed.

ELIGIBILITY:
Inclusion Criteria:

1. With clinical manifestations of influenza.A rapid detection for virus antigen of influenza result is positive.
2. The patients were suffered from influenza within 48 hours.
3. Subjects aged 2 ~14 years old.
4. Before inclusion into the study, The patient's temperature was over 38 ℃.
5. The guardian agreed to participate in this project and signed the informed consent.Patients aged 8 years old or above with their own wishes must be respected.

Exclusion Criteria:

1. Patients with severe or critical illness of influenza.
2. Patients with pneumonia, combined pharyngeal membrane fever, herpetic pharyngitis, suppurative tonsillitis and other diseases.
3. Patients were diagnosed with mycoplasma infection with pharyngeal swab positive or meet the conditions of bacterial infection:White Blood Count(WBC) exceeded 20% of the upper limit of normal range, accompanied by neutrophils increased and serum PCT≥2ug/L, etc.
4. Serum creatinine(SCR) exceeds the upper limit of normal range.Alanine Aminotransferase(ALT) and Aspartate Aminotransferase(AST) exceeded the normal range by more than 2 times.
5. Patients with severe malnutrition, rickets and severe primary diseases of heart, brain, liver, kidney and hematopoietic system.
6. Patients with immunodeficiency or taking glucocorticoid.Patients take other immunosuppressive drugs within the last week.
7. Before be included,patient was taken Oseltamivir or traditional Chinese medicine was used to clear away heat and toxic material within 24 hours.
8. Severely infected persons who must be treated with other antiviral drugs.
9. Allergic to the Reduning injection or Oseltamivir phosphate granules.
10. According to the judgment of the researcher, the patients can cause loss of follow-up should be excluded,such as patients with unstable living environment.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The time of temperature recovery. | If the subject's temperature is less than 37.3℃ and it isn't maintained rise again for 24 hours within 5 days.
  The patients who suffered from influenza were observed their time of temperature recovery .After the first use of the drug,record the time that the patient's temperature dropped to < 37.3℃.The time required for no recurrence within 24 hours.It was the point that evaluated the end of the treatment.

SECONDARY OUTCOMES:
The time when the fever begins to subside | End of day 5.
  The time required for the first drop of body temperature to reach or exceed 0.5℃.
The time of disease to alleviate | End of day 5.
  The symptom score of each symptom after treatment is 0 or mild and lasts for more than 24 hours.The symptom score is recorded daily.
The degree of disease remission | End of day 5.
  According to the"clinical symptom record table", all symptoms were scored.Daily records were recorded to calculate the decrease scores of the total daily symptom score each day.The median time was plotted to calculate Area Under the Curve(AUC) to represent the degree of symptom relief.
The disappearance rate of individual symptoms | End of day 5.
  After medication,patients were asked to evaluate the presence or disappearance of each symptoms (such as fever, headache, body pain, fatigue, pharynx pain, nasal congestion, runny nose, sweating, thirst, cough) of the Influenza.
The rate of negative conversion of Influenza viral | End of day 5.
  The baseline and the end point of treatment were tested for influenza virus in pharyngeal swab.
The number of antipyretic and analgesic drugs used | End of day 5.
  Evaluate the number of combined antipyretic and analgesic drugs used after medication.
The incidence of severe/complications of influenza | End of day 5.
  As the end point of the test,collect data of each participants and calculate the incidence rate of severe/complications of influenza.
Frequency of antipyretic and analgesic drugs used | End of day 5.
  Evaluate the frequency of combined antipyretic and analgesic drugs used after medication.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, Study Principal Investigator, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang S, Xie YM, Wang LX. RDN for the treatment of influenza in children: a randomized, double-blinded, parallel-controlled clinical trial. BMC Complement Med Ther. 2023 Jul 20;23(1):255. doi: 10.1186/s12906-023-04037-1. PMID 37474974